CLINICAL TRIAL: NCT03319030
Title: Evaluating the Impact of Aerobic Exercise in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: Aerobic Exercise in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Aaron Zelikovich, Clinical Research, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: Aerobic Exercise DMD
Record Dates: First submitted 2017-10-09; First posted 2017-10-24 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: exercise; Aerobic Exercise
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Red top blood collection to collect serum microRNA's.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duchenne Muscular Dystrophy (DMD): Enrolls boys with a genetically confirmed diagnosis of DMD.

SUMMARY:
This research study wants to learn more about Duchenne Muscular Dystrophy (DMD) and exercise. Today it is unknown how exercising impacts boys with DMD. The investigators believe that increasing activity and aerobic exercise may help with heart, lung, and muscle function. The investigators are hoping to compare physical strength and blood samples of boys with DMD to see if there are any differences between kids who exercised more as a child versus those who didn't.

DETAILED DESCRIPTION:
Recently, the American Academy of Neurology released new guidelines for children with Duchenne Muscular Dystrophy (DMD) with an updated recommendation to include moderate aerobic exercise. Historically, children with DMD were advised to not exercise as it was thought to accelerate muscle loss. Today, there is new data suggesting that moderate aerobic exercise that does not strain muscle may be beneficial and improve a child's quality of life with regard to heart disease, fatigue, and other factors of overall health. Although it is expected that children who exercise will experience health benefits, there is no scientific evidence indicating a positive or negative effect in a DMD population.

This study is trying to understand the role of aerobic exercise in boys with DMD and how it may impact heart, muscle, and lung function using newly identified biomarkers. The goal is to correlate increased aerobic exercise with improved functional outcomes and changes in biomarkers.

The data collected from this study will allow future development and implementation of an innovative and disease-specific home aerobic exercise program that in the future will be recommended to families of children with DMD.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2-17 years old with a confirmed diagnosis of DMD. Has an appointment in MDA clinic at the Ann & Robert H. Lurie Children's Hospital of Chicago.

Exclusion Criteria:

* Is less than two years old and does not have a confirmed diagnosis of DMD.

Ages: 2 Years to 17 Years | Sex: Male
Age Groups: Child
Gender Based: Yes — X-linked disease. Only males included.
Study Population: The target population is ambulatory and non-ambulatory boys with DMD.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
microRNA levels | Baseline only
  Understanding if there are any differences in microRNA's in boys who are more active versus those who are not.

SECONDARY OUTCOMES:
Physical therapy assessment - 10 meter run test | Baseline only
  Time in seconds that it takes a participant to run 10 meters.
Physical therapy assessment - North Star Ambulatory Assessment | Baseline only
  Comparing a standardized test for ambulatory boys with DMD that gives a score out of 34 total points and microRNA levels.
Physical therapy assessment - time to standing from supine | Baseline only
  Time in seconds that it takes a participant to stand from a supine position.
Cardiac Assessments: Electrocardiogram (ECG) | Baseline only
  Comparing heart rate (BPM), PR interval (msec), QRS (msec), and QT intervals (msec) to microRNA levels.
Cardiac Assessments: Echocardiogram (ECHO) | Baseline only
  Comparing ejection fraction (%) and other Left Ventricle systolic and diastolic metrics (cm) and microRNA levels.
Questionnaire: Pediatric Quality of Life: Neuromuscular module | Baseline only
  To see if there is any correlation between Quality of Life scores (range from 0 to 100) and microRNA levels. Increased scores indicate a higher quality of life.
Questionnaire: Physical Function Survey | Baseline only
  To see if there is any correlation between scores of functional ability (with a range from 0 to 106) and microRNA levels. Higher physical function function scores indicate increased strength.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Zelikovich, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guiraud S, Aartsma-Rus A, Vieira NM, Davies KE, van Ommen GJ, Kunkel LM. The Pathogenesis and Therapy of Muscular Dystrophies. Annu Rev Genomics Hum Genet. 2015;16:281-308. doi: 10.1146/annurev-genom-090314-025003. Epub 2015 Jun 4. PMID 26048046
- [Background] Flanigan KM, Ceco E, Lamar KM, Kaminoh Y, Dunn DM, Mendell JR, King WM, Pestronk A, Florence JM, Mathews KD, Finkel RS, Swoboda KJ, Gappmaier E, Howard MT, Day JW, McDonald C, McNally EM, Weiss RB; United Dystrophinopathy Project. LTBP4 genotype predicts age of ambulatory loss in Duchenne muscular dystrophy. Ann Neurol. 2013 Apr;73(4):481-8. doi: 10.1002/ana.23819. Epub 2013 Feb 20. PMID 23440719
- [Background] Hathout Y, Marathi RL, Rayavarapu S, Zhang A, Brown KJ, Seol H, Gordish-Dressman H, Cirak S, Bello L, Nagaraju K, Partridge T, Hoffman EP, Takeda S, Mah JK, Henricson E, McDonald C. Discovery of serum protein biomarkers in the mdx mouse model and cross-species comparison to Duchenne muscular dystrophy patients. Hum Mol Genet. 2014 Dec 15;23(24):6458-69. doi: 10.1093/hmg/ddu366. Epub 2014 Jul 15. PMID 25027324
- [Background] Giordani L, Sandona M, Rotini A, Puri PL, Consalvi S, Saccone V. Muscle-specific microRNAs as biomarkers of Duchenne Muscular Dystrophy progression and response to therapies. Rare Dis. 2014 Dec 1;2(1):e974969. doi: 10.4161/21675511.2014.974969. eCollection 2014. PMID 26942105
- [Background] Cacchiarelli D, Legnini I, Martone J, Cazzella V, D'Amico A, Bertini E, Bozzoni I. miRNAs as serum biomarkers for Duchenne muscular dystrophy. EMBO Mol Med. 2011 May;3(5):258-65. doi: 10.1002/emmm.201100133. Epub 2011 Mar 21. PMID 21425469
- [Background] Baggish AL, Park J, Min PK, Isaacs S, Parker BA, Thompson PD, Troyanos C, D'Hemecourt P, Dyer S, Thiel M, Hale A, Chan SY. Rapid upregulation and clearance of distinct circulating microRNAs after prolonged aerobic exercise. J Appl Physiol (1985). 2014 Mar 1;116(5):522-31. doi: 10.1152/japplphysiol.01141.2013. Epub 2014 Jan 16. PMID 24436293
- [Derived] Quattrocelli M, Zelikovich AS, Jiang Z, Peek CB, Demonbreun AR, Kuntz NL, Barish GD, Haldar SM, Bass J, McNally EM. Pulsed glucocorticoids enhance dystrophic muscle performance through epigenetic-metabolic reprogramming. JCI Insight. 2019 Dec 19;4(24):e132402. doi: 10.1172/jci.insight.132402. PMID 31852847